CLINICAL TRIAL: NCT03565562
Title: Preventing Psychological Distress and Suicidal Behaviours: a Web-based and Mobile Suicide Prevention Intervention in the General Population
Acronym: PRINTEMPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: National Agency of Public Health (Other); Centre Collaborateur OMS pour la recherche et la formation en santé mentale (Unknown); Institut de Recherche en Santé Publique, France (Other); UMR INSERM 1246 - SPHERE MethodS in Patients-centered outcomes and HEalth ResEarch (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C 15-45
Record Dates: First submitted 2018-04-20; First posted 2018-06-21 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2019-12

CONDITIONS: Suicide and Depression; Psychological Distress; Anxiety Disorders; Local Authorities Promotion
Keywords: Health promotion; Local authorities involvement; Suicide and attempted suicide; Primary prevention; Psychological Distress
MeSH Terms: conditions — Suicide; Depression; Anxiety Disorders; Suicide, Attempted

STUDY DESIGN:
Intervention Model Description: cluster randomized, open parallel groups , controlled intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (No Intervention): Local authorities allocated to this group won't implement any promotion of the e-health tool for the 12 first months. Free access to StopBlues.
- Group experimental 1 promotion (Active Comparator): Local authorities allocated to this group will have to implement the promotion of the e-health tool: the promotion at the local authority level. They will promote the e-health tool using their usual communication methods (local newspapers, local website, bulletin and billboards, posters in the local shops and in the bus stops…). Free access to StopBlues.
  Interventions: Other: Promotion of the e-health tool by local authorities
- Group experimental 2 promotion (Active Comparator): Local authorities allocated to this group will have to implement promotion of the e-health tool: the promotion at local authority and GPs' waiting room level. Local authorities will promote the e-health tool using their usual communication methods (local newspapers, local website, bulletin and billboards, posters in the local shops and in the bus stops...). (similarly to group experimental1) as well as leaflets and posters in GPs' waiting room. Free access to StopBlues.
  Interventions: Other: Promotion of the e-health tool by local authorities; Other: Promotion of the e-health tool by local authorities and GPs

INTERVENTIONS:
Other: Promotion of the e-health tool by local authorities — Local authorities participating in the trial will select a referent person who will be in charge of the implementation and follow-up of the promotion. A promotion toolkit with recommendations, posters, web banners, leaflets and ready-made messages and press articles will be provided to the local authorities.
  Other Names: StopBlues
  Arms: Group experimental 1 promotion; Group experimental 2 promotion
Other: Promotion of the e-health tool by local authorities and GPs — In those local authorities, GPs will participate passively to the promotion of the e-health tool, by providing posters and leaflets in their waiting rooms.
  Other Names: StopBlues
  Arms: Group experimental 2 promotion

SUMMARY:
An interventional research study will be undertaken to assess the effectiveness of the promotion at the local level of an e-health tool for suicide and psychological distress prevention (the StopBlues application and website). This trial is a cluster-randomized, parallel group, controlled intervention study with local authorities as the unit of randomization. Local authorities will be randomly assigned to one of the following three arms: local authorities not promoting the e-health tool (control group); local authorities promoting the e-health tool without general practitioners (GPs) involvement; local authorities promoting the e-health tool including GPs' waiting room. The trial will last 24 months and after a 12-month post-randomization period, local authorities from the control group will be allowed for a further 12-month period to launch their promotional campaign supported by the research team through regular contacts and additional technical and financial resources (intensively sustained promotion). This will facilitate the recruitment of clusters as well as their adherence to the intervention during the first 12-month period. The main criterion will be the number of suicidal acts at nine months. Data will be collected both at the local authority level and at the individual e-health tool user level.

DETAILED DESCRIPTION:
* Context France is one of the Western European countries most affected by suicide, which is associated with a high societal cost. Recently, a European project aiming to develop best practice for suicide prevention has recommended the development of web-based interventions and the French national plan for actions against suicide has supported the development of reference websites for suicide prevention. However, web-based interventions should be associated with effective promotional efforts to ensure awareness but also to improve receptiveness among and around those who could benefit from such a resource. Previous work has shown that local authorities are appropriate actors for promoting prevention measures against suicide and that 20% of individuals attempting suicide visit their GP the day before their attempt.
* Research objectives The primary objective of our trial is to assess the effectiveness of the tailored promotion at local level of an e-health tool and to compare the effectiveness at 12 months of two types of local promotion (with or without involving GPs' waiting room) on suicidal acts. The secondary objectives are to assess the cost-effectiveness and to run a budgetary impact analysis of the intervention. Moreover, our secondary objectives are to assess the effectiveness of the promotion on the intensity of utilization of StopBlues by the three types of users (living in a city without promotion or with promotion or reinforced promotion), on their help-seeking behavior, on their implementation of supportive activities into their daily life and on the evolution of users level of psychological impairment. An additional form of promotion (intensively sustained promotion) will be implemented after 12 months in the control group and evaluated using the same primary outcome measure. In parallel, the long-term effectiveness of the two main types of local promotion (with or without a passive involvement of GPs through their waiting room) will also be assessed.
* Methodology The detailed content of the e-health tool and the promotional tools to be made available to local authorities and GPs was determined through literature reviews and focus groups with experts and users.

A cluster-randomized, parallel group, controlled intervention study with local authorities as the unit of randomization will be set up. Local authorities can either be cities or a grouping of cities ("communauté de communes"), based on the local health governance of each area. If several adjacent local authorities volunteer individually to participate in the trial, they will be considered as a unique local authority. Volunteer local authorities will be randomly assigned to one of the following three arms: those not promoting the e-health tool (control group); those promoting the e-health tool without involving GPs' waiting rooms; those promoting the e-health tool involving GPs' waiting rooms.

The trial will last 24 months and local authorities will be able to switch arm if they so wish after 12 months and launch an 'intensively sustained promotion'. This will facilitate recruitment of local authorities as well as their adherence to the intervention. Data will be collected both at the local authority level and at the individual user level.

• Expected results The investigators anticipate that the promotion of the e-health intervention will lead to a greater difference in the number of suicidal acts in the local authorities where it is implemented over the trial period. Furthermore, it should also result in a higher reduction of psychological distress and in an increased intensity and length of use of the e-health tool. The promotion may also lead members of the population with moderate level of psychological distress, who may not otherwise be seeking help, to access the e-health tool and should also facilitate help-seeking behaviors and implementation of supportive activities into their daily life. The intensively sustained promotion should lead to higher rates of connexion and by then to a higher reduction of psychological distress and in an increased intensity and length of use of the e-health tool.

Moreover, this project will give information on the relevance of our promotion model for primary prevention of psychological distress. Indeed, if the findings are satisfactory, this model and the formalized networks for promotion within local authorities may facilitate development of additional primary prevention measures both for mental disorders and other health issues.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* living in one of the 42 french local authority participating to the trial
* volunteer
* access to internet (smartphone/tablet/computer)

Exclusion Criteria:

* <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100000 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Number of suicides - Short term | At month 9
  The number of completed suicides will be extracted from the database of the Epidemiology center on medical causes of deaths (CépiDc) for each local authority participating.
Number of suicide attempts - Short term | At month 9
  The number of attempted suicides will be extracted from the national database of public and private hospital admissions (PMSI-MCO) and the national emergency database (Oscour).

SECONDARY OUTCOMES:
Number of suicides - Long term | At the end of the trial (month 18)
  The number of completed suicides will be extracted from the database of the Epidemiology center on medical causes of deaths (CépiDc) for each local authority participating.
Number of suicide attempts - Long term | At the end of the trial (month 18)
  The number of attempted suicides will be extracted from the national database of public and private hospital admissions (PMSI-MCO) and the national emergency database (Oscour).
Costs | At 9 months and at the end of the trial (month 18)
  Fixed costs for the development of the intervention including promotions tools, semi-fixed costs for the implementation of the program by local authorities and GPs, costs of suicidal acts.
Level of health-related quality of life and associated utility of StopBlues users | At registration, and 1, 2, 3, 6, 12 and 18 months after
  Collected through self-assessment at the user level with the quality of life questionnaire Short Form-12 (SF-12).
Level of psychological pain of StopBlues users | At registration, and then at 1, 2, 3, 6, 12 and 18 months
  Collected through self-assessment at the user level with the 12-item General Health Questionnaire (GHQ-12).
Level of depression of StopBlues users | At registration, and then at 1, 2, 3, 6, 12 and 18 months
  Collected through self-assessment at the user level with the Patient Health Questionnaire (PHQ-9)
Level of anxiety of StopBlues users | At registration, and then at 1, 2, 3, 6, 12 and 18 months
  Collected through self-assessment at the user level with the General Anxiety Disorder questionnaire (GAD-7).
Level of suicidal risk of StopBlues users | At first filling and 1, 2, 3, 6, 12 and 18 months after
  Collected through self-assessment at the user level with the 6 questions on the suicidal risk of the Mini International Neuropsychiatric Interview-Simplified (MINI-S). The MINI-S is not available at registration, it will be triggered when results to GHQ-12, PHQ-9 and/or GAD-7 are considered showing a suicidal risk for the user.
Help-seeking behaviors and implementation of supportive activities into daily life of StopBlues users | At registration, and 1, 2, 3, 6, 12 and 18 months after
  Collected through self-assessment at the user level with an ad hoc questionnaire adapted from the general health-seeking questionnaire (GHSQ).
Level of depression (for StopBlues users coming for a relative) | At registration
  Collected at the user level with the Montgomery-Asberg Depression Scale (MADRS). It has 10 questions, quoted from 0 to 6.
Intention to seek help of StopBlues users | At registration for users coming for a relative, and at registration and 1, 2, 3, 6, 12 and 18 months after for users coming for themselves
  French traduction of the first question of the General Help-Seeking Questionnaire -Original Version (GHSQ).
Intensity of the participation to the application and website | At month 9 and 18 (end of the trial)
  Number of downloads and connections for each zip codes of local authorities included in the trial.
Length of use to the application and website | At month 9 and 18 (end of the trial)
  Time-lapse between the inscription and the last connection to the application or website.
Proportion of StopBlues users who came to know the e-health tool through the different communication channels | At registration
  Collected at the user level with a specific question: "How did you get to know about the StopBlues program?" .
  1/ By public display 2/ In public places (employment center, library ...) 3/ On my city website 4/ By the press 5/ Through social networks 6/ At merchants 7/ At my pharmacist 8/ At my GP 9/ At another health professional (physiotherapist, medical specialist ...) 10/Through relationships (friends, families, neighbors ...) 11/ Other
Proportion of StopBlues users who came for a relative | At registration
  The proportion of users who subscribed for a relative and not for themselves.
StopBlues users with a safety plan | At month 9 and 18 (end of the trial)
  The proportion of users who filled up a safety plan.

CONTACTS AND LOCATIONS:
Overall Officials: Karine Chevreul, MD, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Faculté de Médecine Paris Diderot Paris 7, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bertolote J, Fleischmann A. A global perspective on the magnitude of suicide mortality. The Oxford Textbook of Suicidology and Suicide Prevention: A Global Perspective. Oxford: Oxford University Press. Wasserman D., Wasserman C.; 2009. p. 91 98.
- [Background] Marie-Claude Mouquet, Bellamy V. Suicides et tentatives de suicide en France. Etude et Résultats. Mai 2006;(488).
- [Background] O'Dea D, Tucker S. The cost of suicide to society. Wellington: Ministry of Health. 2005.
- [Background] Kennelly B. The economic cost of suicide in Ireland. Crisis. 2007;28(2):89-94. doi: 10.1027/0227-5910.28.2.89. PMID 17722690
- [Background] du Roscoat E, Beck F. Efficient interventions on suicide prevention: a literature review. Rev Epidemiol Sante Publique. 2013 Aug;61(4):363-74. doi: 10.1016/j.respe.2013.01.099. Epub 2013 Jul 10. PMID 23849295
- [Background] Warnet S. [New national program for the prevention of suicide]. Rev Infirm. 2011 Nov;(175):4. No abstract available. French. PMID 22206200
- [Background] Ministère des Affaires Sociales et de la Santé. Décret n° 2013-809 du 9 septembre 2013 portant création de l'Observatoire National du Suicide. 2013
- [Background] Atkinson NL, Saperstein SL, Pleis J. Using the internet for health-related activities: findings from a national probability sample. J Med Internet Res. 2009 Feb 20;11(1):e4. doi: 10.2196/jmir.1035. PMID 19275980
- [Background] Dickerson S, Reinhart AM, Feeley TH, Bidani R, Rich E, Garg VK, Hershey CO. Patient Internet use for health information at three urban primary care clinics. J Am Med Inform Assoc. 2004 Nov-Dec;11(6):499-504. doi: 10.1197/jamia.M1460. Epub 2004 Aug 6. PMID 15298993
- [Background] Haga SM, Drozd F, Brendryen H, Slinning K. Mamma mia: a feasibility study of a web-based intervention to reduce the risk of postpartum depression and enhance subjective well-being. JMIR Res Protoc. 2013 Aug 12;2(2):e29. doi: 10.2196/resprot.2659. PMID 23939459
- [Background] Monshat K, Vella-Brodrick D, Burns J, Herrman H. Mental health promotion in the Internet age: a consultation with Australian young people to inform the design of an online mindfulness training programme. Health Promot Int. 2012 Jun;27(2):177-86. doi: 10.1093/heapro/dar017. Epub 2011 Mar 11. PMID 21398335
- [Background] Allen J, Mohatt G, Fok CC, Henry D; People Awakening Team. Suicide prevention as a community development process: understanding circumpolar youth suicide prevention through community level outcomes. Int J Circumpolar Health. 2009 Jun;68(3):274-91. doi: 10.3402/ijch.v68i3.18328. PMID 19705659
- [Background] Bean G, Baber KM. Connect: an effective community-based youth suicide prevention program. Suicide Life Threat Behav. 2011 Feb;41(1):87-97. doi: 10.1111/j.1943-278X.2010.00006.x. Epub 2011 Jan 24. PMID 21309827
- [Background] Ono Y, Sakai A, Otsuka K, Uda H, Oyama H, Ishizuka N, Awata S, Ishida Y, Iwasa H, Kamei Y, Motohashi Y, Nakamura J, Nishi N, Watanabe N, Yotsumoto T, Nakagawa A, Suzuki Y, Tajima M, Tanaka E, Sakai H, Yonemoto N. Effectiveness of a multimodal community intervention program to prevent suicide and suicide attempts: a quasi-experimental study. PLoS One. 2013 Oct 9;8(10):e74902. doi: 10.1371/journal.pone.0074902. eCollection 2013. PMID 24130673
- [Background] Pearson A, Saini P, Da Cruz D, Miles C, While D, Swinson N, Williams A, Shaw J, Appleby L, Kapur N. Primary care contact prior to suicide in individuals with mental illness. Br J Gen Pract. 2009 Nov;59(568):825-32. doi: 10.3399/bjgp09X472881. PMID 19861027
- [Background] Hegerl U, Althaus D, Schmidtke A, Niklewski G. The alliance against depression: 2-year evaluation of a community-based intervention to reduce suicidality. Psychol Med. 2006 Sep;36(9):1225-33. doi: 10.1017/S003329170600780X. Epub 2006 May 17. PMID 16707028
- [Background] Chabaud F, Debarre J, Serazin C, Bouet R, Vaiva G, Roelandt JL. [Study of population profiles in relation to the level of suicide risk in France: Study "Mental health in the general population"]. Encephale. 2010;36(3 Suppl):33-8. doi: 10.1016/S0013-7006(10)70016-6. French. PMID 20813223
- [Background] Campbell MK, Piaggio G, Elbourne DR, Altman DG; CONSORT Group. Consort 2010 statement: extension to cluster randomised trials. BMJ. 2012 Sep 4;345:e5661. doi: 10.1136/bmj.e5661. No abstract available. PMID 22951546
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Background] Schmidtke A, Bille-Brahe U, DeLeo D, Kerkhof A, Bjerke T, Crepet P, Haring C, Hawton K, Lonnqvist J, Michel K, Pommereau X, Querejeta I, Phillipe I, Salander-Renberg E, Temesvary B, Wasserman D, Fricke S, Weinacker B, Sampaio-Faria JG. Attempted suicide in Europe: rates, trends and sociodemographic characteristics of suicide attempters during the period 1989-1992. Results of the WHO/EURO Multicentre Study on Parasuicide. Acta Psychiatr Scand. 1996 May;93(5):327-38. doi: 10.1111/j.1600-0447.1996.tb10656.x. PMID 8792901
- [Background] Réseau OSCOUR® / Surveillance syndromique - SurSaUD® / Veille et alerte / Dossiers thématiques / Accueil [Internet]. Disponible sur: http://www.invs.sante.fr/Dossiers-thematiques/Veille-et-alerte/Surveillance-syndromique-SurSaUD-R/Reseau-OSCOUR-R
- [Background] HAS. Choix méthodologiques pour l'évaluation économique à la HAS. 2011
- [Derived] Turmaine K, Dumas A, Chevreul K; PRINTEMPS Consortium. Conditions for the Successful Integration of an eHealth Tool "StopBlues" Into Community-Based Interventions in France: Results From a Multiple Correspondence Analysis. J Med Internet Res. 2022 Apr 22;24(4):e30218. doi: 10.2196/30218. PMID 35451977
- [Derived] Gandre C, Le Jeannic A, Vinet MA, Turmaine K, Courtet P, Roelandt JL, Vaiva G, Giraudeau B, Alberti C, Chevreul K. The PRINTEMPS study: protocol of a cluster-randomized controlled trial of the local promotion of a smartphone application and associated website for the prevention of suicidal behaviors in the adult general population in France. Trials. 2020 Jun 22;21(1):553. doi: 10.1186/s13063-020-04464-2. PMID 32571432